CLINICAL TRIAL: NCT05525221
Title: Societal Merit of Intervention on Hearing Loss Evaluation - Investigating the Impact of (Waiting for) Cochlear Implantation in People With Severe to Profound Sensorineural Hearing Loss on Societal Related Outcomes.
Brief Title: Societal Merit of Intervention on Hearing Loss Evaluation
Acronym: SMILE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-6057
Record Dates: First submitted 2022-08-25; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Bilateral; Hearing Loss, Adult-Onset; Hearing Loss, Bilateral Sensorineural, Progressive
Keywords: Cochlear Implantation
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral; Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The primary objective of this study is to determine the (long term) effect of intervention with a CI in adult participants with progressive postlingual moderate/severe-to-profound sensorineural hearing loss on societal related outcomes (participation; communication profile; autonomy; cognition; listening effort; work; productivity loss; income; medical consumption; third party quality of life; quality of life, and capability).

The secondary objective is to determine the effect of CI waiting time between referral and CI surgery on the same societal related outcomes, in the adults with postlingual moderate/severe-to-profound sensorineural hearing loss.

DETAILED DESCRIPTION:
Cochlear implantation (CI) is a surgical intervention to improve the hearing of patients with profound hearing loss. Due to the improvements in CI-technology and knowledge regarding surgery and CI fitting, speech recognition with CI has improved over the past decades. This has led to relaxation of the audiological implantation criteria. Whereas CI was initially indicated for patients with total deafness, currently also patients with moderate/severe-to-profound hearing loss are eligible for CI.

Moderate/severe-to-profound hearing loss has a negative effect on the patients' functioning. Because often hearing loss in adults is progressive, resulting in a decline in speech recognition, the disability might progress during this waiting time to a state in which societal participation can become even more difficult: the hearing loss might affect social participation, autonomy, work/occupational status and quality of life. However empirical data on this is not yet available. Timely intervention, like cochlear implantation may prevent societal drop out.

The societal impact of cochlear implantation for patients who are (currently) eligible for CI is unknown. It is imperative to obtain this data in order to secure treatment for those who need it. This multicenter cohort observational study is set up to investigate the impact of moderate/severe-to-profound hearing loss on societal related outcomes, defined as participation; communication profile; autonomy; cognition; listening effort; work; productivity loss; income; medical consumption; third party quality of life; quality of life, and capability. The primary aim is to investigate the effect of hearing rehabilitation with cochlear implantation on these societal related outcomes.

Castoredc (Castor electronic data capture) will be used for capturing research data. Questionnaires will be constructed in castors' online survey service and administered to participants online.

IBM SPSS Statistics and R studio software will be used for the statistical analysis. Descriptive analysis will be conducted to assess the baseline characteristics and the continuous variables will be summarized with mean ± SD or median (interquartile range) (if not normally distributed) and categorical variables with percentage (numbers). The statistical analysis for the primary objective, the differences in baseline(T0) and T2/T3/T4 for the primary outcome variables, we will use general linear models with the outcome (differences) as independent variable. To investigate the complete pattern in time of the effects we will use mixed models, in which time is an additional explanatory categorical variable. For the secondary objective the effect between baseline(T0) and T1, short before CI surgery will be investigated. General linear models with the outcome (differences) as independent variable.

ELIGIBILITY:
Inclusion Criteria:

* Adults (potentially) eligible for CI according to the Dutch quality standard for CI (Veldnorm CI 2013) and willing to participate. Participants are divided in 2 age categories (under and over 65 years old)

Exclusion Criteria:

* People with a complex syndrome with multiple problems.
* Incapable of performing paid or unpaid labor, due to non-hearing related factors
* Prelingual onset of deafness.
* Children 0 - 18 years old.
* Non-native Dutch speakers.
* Patients suffering from a psychiatric disorder
* Any condition that may hamper a complete insertion of the electrode array or a normal rehabilitation with the cochlear implant (severe otosclerosis or neurologic deficits)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with moderate-severe to profound hearing loss who are referred to a tertiary hospital for potentially receiving a cochlear implant.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2020-06-29 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Participation | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  Sub-scales ('family role', 'Social life and relationships' and 'work and education') of The Impact on Participation and Autonomy questionnaire (IPA).There are 4 response options for each of the 32 items about participation and autonomy. These response options range from 'very good' (score=0) to 'bad' (score =4). There are 3 response options for the items about problem experiences. These range from 'no problem' (score=0) to 'big problem'(score=2). The scores of the 32 options will be summarized per sub-scale.

SECONDARY OUTCOMES:
Change in Autonomy | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  Sub-scales ('Autonomy indoors' and 'Autonomy outdoors') of The Impact on Participation and Autonomy questionnaire (IPA)
Change in Communication profile | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  Amsterdam questionnaire for Hearing and Work. Subscales derived from the Communication Profile for Hearing Impaired (CPHI) questionnaire: 'use of communication strategies' consists of: Maladaptive Behaviors; Verbal Strategies and Non-verbal Strategies
  'Personal adjustment to hearing impairment' consists of: Self-acceptance; Acceptance of loss; Stress an Withdrawal.
Change in Work experience and status | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  Amsterdam questionnaire for Hearing and Work.Three scales: Subscales originated from the Vragenlijst Beleving en Beoordeling van de Arbeid (VBBA) [Questionnaire on Experience and appreciation of labor]. Subscale are: participation ['inspraak'], relationship with co-workers [relatie met collega's], Need for recovery [herstelbehoefte].
Change in Work capabilities | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  List Work Capabilities. Sum score of total capability set for work. Because people want to achieve personal important goals and values in their work the List Work Capabilities (LWC) measures sustainable employability based on seven important labor values that are identified in previous studies. The scope of the LWC is not on health or broader economic indicators such as (sick leave) costs and benefits, rather it investigates values that the employee can realize in their specific work context.
Change in Productivity Costs Questionnaire | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  The Productivity Cost Questionnaire (PCQ). Health problems often have a negative impact on the capacity for patients to maintain paid or unpaid work. From a societal perspective this productivity loss has an impact and should therefore be measured in a validated manner. The PCQ consists of 3 modules: absenteeism, presenteeism and Productivity loss at unpaid work.
Change in Medical Consumption Questionnaire | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  In economic evaluations it is important to include direct costs within the healthcare system. These costs are directly related to prevention, diagnostics, therapy, rehabilitation and care of a disease or disorder. Patients are involved in their resource (health care) consumption and are therefore a reliable source of information. The consumption of health care in a variety of costs components will be investigate by the use of the medical consumption questionnaire.
Change in Capability | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  ICECAP-A. The ICECAP-A is a measure of capability for adults. The ICECAP focuses on wellbeing defined in a broader sense, rather than health. It is a questionnaire that comprises 5 attributes. Attachment, Stability, Achievement, Enjoyment, Autonomy.
Change in Generic Quality of Life (EQ5D-5L) | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  EuroQol five-dimension scale questionnaire (EQ5D-5L)
Change in Generic Quality of Life (HUI-3) | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  Health Utility Index Mark 3 (HUI-3)
Change in Third Party Hearing loss related quality of life measured by Hearing Impairment Impact-Significant Other Profile (HII-SOP). | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  The HII-SOP is a 20-item scale with three subscales: 1) Emotions that arise when having a spouse with hearing loss as well as the impact of the hearing loss on the marital relationship, 2) The impact of the hearing loss on the social life of the spouse, and 3) the communication strategies used by the spouse
Change in Disease specific Quality of Life measured by Nijmegen Cochlear Implant Questionnaire (NCIQ) | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  Comprising of subdomains; Basic sound perception; Advanced sound perception; Speech production; Self-esteem; Activity limitations; Social interaction.
Change in Income (source) | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  Questions investigating the sources of income and selecting income brackets.
Change in Cognition | Once between study inclusion and surgery (pre-operative), 1 year post surgery, and (if participant is over 65 years old) 2 years post surgery.
  Repeatable Battery for the Assessment of Neuropsychological Status for Hearing impaired (RBANS-H).This cognitive test assesses five cognitive domains; Immediate Memory, Visuospatial/constructional, Language, Attention and Delayed Memory. Within these domains there are 12 subtests. Subdomain scores and total scores will be calculated at various time points. This tests will be conducted in participants included in one of the centers.
Change in Listening effort | 4 weeks after surgery and 1 year after surgery.
  Listening effort will be assessed in a sub-population of participants under 65 by using pupillometry
Change in Linguistic skills by Vocabulary test | Once between inclusion and surgery.
  Adaptive Vocabulary test STAIRS4WORDS developed by the Max Planck Institute for Psycholinguistics.
Change in Tinnitus | T0 (baseline), T1 (pre-operative, if waiting time > 6 months), T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  Measured by the THI (Tinnitus Handicap Inventory)
Change in quality of life score post-intervention | T2 (1 year post CI surgery), T3 (2 years post CI surgery), T4 (3 years post CI surgery)
  Measured by The Glasgow Benefit Inventory (GBI)

OTHER OUTCOMES:
Change in Audiological outcomes Tone thresholds | Pre-surgery and 1 year post-surgery
  Pure tone Thresholds air and bone conduction (aided and un-aided) on frequency that are considered clinically relevant by the conducting audiologist.
Change in Audiological outcomes speech perception score unaided by using NVA lists and CVC words/phonemes. | Pre-surgery and 1 year post-surgery
  Speech perception unaided at 85, 75 and 65 dBSPL
Change in Audiological outcomes speech perception score aided by using NVA lists and CVC words/phonemes. | Pre-surgery and 1 year post-surgery
  Speech perception aided at 75, 65 and 55 dBSPL
Change in Audiological outcomes - speech perception score aided free field by using NVA lists and CVC words/phonemes. | Pre-surgery and 1 year post-surgery
  Speech perception aided in free field at 65 and 55 dBSPL

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Mylanus, Study Director — Radboud University Medical Center
Locations (5):
- Netherlands (5):
  - Radboudumc, Nijmegen, Gelderland
  - Maastricht UMC+, Maastricht, Limburg
  - Amsterdam UMC, Amsterdam, North Holland
  - Leids UMC, Leiden, South Holland
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] Beckers L, Nijmeijer H, Mylanus E, Huinck W. Investigating the association between pre-implantation cognitive performance and one-year post-implantation speech perception outcomes in adult cochlear implant recipients using the repeatable battery for the assessment of neuropsychological status for hearing impaired individuals (RBANS-H). Cochlear Implants Int. 2025 Dec 22:1-12. doi: 10.1080/14670100.2025.2601419. Online ahead of print. PMID 41431315
- [Derived] Nijmeijer HGB, Philpott N, van der Wilt GJ, Donders ART, George E, Boerboom R, Frijns JHM, Kaandorp M, Huinck WJ, Mylanus EAM. Changes in participatory and societal outcomes during the waiting period for cochlear implantation - an observational study. Eur Arch Otorhinolaryngol. 2025 Feb;282(2):753-764. doi: 10.1007/s00405-024-08981-7. Epub 2024 Sep 26. PMID 39327291
- [Derived] Nijmeijer HGB, Huinck WJ, Kramer SE, Donders ART, van der Wilt GJ, Mylanus EAM. Changes on clinical and participatory outcomes in people with severe-to-profound hearing loss after cochlear implantation: protocol of a multicentre prospective observational cohort study - Societal Merit of Intervention on Hearing Loss Evaluation (SMILE). BMJ Open. 2023 Jun 27;13(6):e072689. doi: 10.1136/bmjopen-2023-072689. PMID 37369408